CLINICAL TRIAL: NCT02496624
Title: Cone-beam Computed Tomography (CT) Guided Microcoil Localization of Pulmonary Nodules During Video Assisted Thoracic Surgery(VATS)
Brief Title: Cone-beam CT Guided Microcoil Localization of Pulmonary Nodules During Video Assisted Thoracic Surgery(VATS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14-7395
Record Dates: First submitted 2015-07-06; First posted 2015-07-14 (Estimated); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lung cancer (Other)
  Interventions: Other: Cone Beam CT localization and placement of microcoil

INTERVENTIONS:
Other: Cone Beam CT localization and placement of microcoil — Cone Beam CT localization and placement of microcoil

SUMMARY:
The Guided Therapeutics (GTx) program at the University Health Network is a network of clinicians, scientists, and engineers focused on the development and translation of image-guided technologies focused on minimally-invasive, adaptive therapies. Technologies developed within the GTx program include a portable intra-operative cone-beam CT (in collaboration with Siemens) that has been evaluated in clinical trials for head and neck surgery. The intraoperative imaging has been integrated with tracking and navigational tools and optical imaging to provide a general "surgical dashboard" that is used to improve the accuracy of surgical resection.

A recent addition to the GTx program is the development of the GTx OR, located within the general operating room of the Toronto General Hospital. The GTx OR houses 2 complimentary advance technologies: the Siemens Zeego and the Siemens Somotom Flash CT. The dual-energy Somatom Flash provides a "gold-standard" in CT imaging, while the Zeego provides excellent 3D Cone-beam CT with robotic placement for flexible integration within the operating environment. Together, the integration of these 2 components into a single OR enables critical evaluation of the limits of CT imaging technology for surgical guidance.

This study will be conducted using solely the Cone-beam CT (Zeego) for percutaneous placement and localization of markers for resection of small pulmonary nodules during VATS.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient age 18 and older with lung nodules who are candidates for microcoil localization prior to VATS wedge resection

Exclusion Criteria:

* Patients that are unable to give informed consent
* Patients that are unable to tolerate general anesthesia
* Patients who are pregnant or patients that believe they are pregnant
* Patients with implantable devices susceptible to Radio Frequency (RF) fields
* Severely obese patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-06; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Radiation Exposure | 4 years
  Will determine how much radiation the patient receives via CT report
Length of time to perform procedure | 4 years
  Will time the procedure in order to determine procedure length

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada